CLINICAL TRIAL: NCT06631625
Title: Effect of Dexmedetomidine/Lidocaine, Ketamine/Lidocaine and Lidocaine Alone on Proinflammatory Cytokines in Pelvi-abdominal Cancer Surgeries: Randomised Prospective Study
Brief Title: Effect of Addition of Dexmedetomidine or Ketamine to Intravenous Infusion of Lidocaine on Proinflammatory Cytokines in Pelvi-abdominal Cancer Surgeries.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Bassem Emad, Assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0202037
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Pelvic Cancer; Abdominal Cancer; Surgery; Proinflammatory Cytokines
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group L receiving intravenous lidocaine infusion only (Experimental): Patients will receive 1.5mg /kg lidocaine 2%; intravenously as a bolus dose then 1.5mg/kg/hr lidocaine infusion using a 50cc syringe pump intra-operatively.
  Interventions: Drug: Lidocaine Intravenous Infusion
- Group LK receiving lidocaine and ketamine infusion (Experimental): Patients will receive same infusion regimen of lidocaine 2%; as in group L plus 0.35 mg/kg ketamine intravenously as a bolus dose, followed by intravenous infusion of 0.2 mg/kg/h using a 50cc syringe pump intra- operatively.
  Interventions: Drug: Lidocaine and ketamine
- Group LD receiving lidocaine and dexmedetomidine infusion (Experimental): Patients will receive same infusion regimen of lidocaine 2%; as in group L plus 0.5 μg/kg dexmedetomidine intravenously as a bolus dose, followed by intravenous infusion of 0.4 μg/kg/h using a 50cc syringe pump intra-operatively.
  Interventions: Drug: lidocaine and dexmedetomidine infusion

INTERVENTIONS:
Drug: Lidocaine Intravenous Infusion — Patients will receive 1.5mg /kg lidocaine 2%; intravenously as a bolus dose then 1.5mg/kg/hr lidocaine infusion using a 50cc syringe pump intra-operatively.
  Arms: Group L receiving intravenous lidocaine infusion only
Drug: Lidocaine and ketamine — Patients will receive same infusion regimen of lidocaine 2%; as in group L plus 0.35 mg/kg ketamine intravenously as a bolus dose, followed by intravenous infusion of 0.2 mg/kg/h using a 50cc syringe pump intra- operatively.
  Arms: Group LK receiving lidocaine and ketamine infusion
Drug: lidocaine and dexmedetomidine infusion — Patients will receive same infusion regimen of lidocaine 2%; as in group L plus 0.5 μg/kg dexmedetomidine intravenously as a bolus dose, followed by intravenous infusion of 0.4 μg/kg/h using a 50cc syringe pump intra-operatively.
  Arms: Group LD receiving lidocaine and dexmedetomidine infusion

SUMMARY:
The investigators hypothesize that effect of addition of dexmedetomidine or ketamine by IV infusion to lidocaine infusion may be more beneficial than lidocaine infusion alone on proinflammatory cytokines (IL-1, IL-6 and TNFα), and postoperative pain relief and decreased opioid consumption, reduced Length of stay.

DETAILED DESCRIPTION:
45 female patients of American Society of Anesthesiologists (ASA) physical status I or II, aged (40-70) years admitted to department of obstetrics and gynecology, El shatby University Hospital and scheduled for elective pelvi- abdominal cancer surgery. Patients will be randomly allocated using a computer generated random table (Graphpad Software, Inc, La Jolla, CA) and an allocation ratio of 1:1 using a sealed envelope method to one of three groups. The envelope will be opened by an observer not involved in the study. Patients will be divided into three equal groups. Group L (n=15): Patients will receive 1.5mg /kg lidocaine 2%; intravenously as a bolus dose then 1.5mg/kg/hr lidocaine infusion using a 50cc syringe pump intra-operatively. Group LK (n=15): Patients will receive same infusion regimen of lidocaine 2%; as in group L plus 0.35 mg/kg ketamine intravenously as a bolus dose, followed by intravenous infusion of 0.2 mg/kg/h using a 50cc syringe pump intra- operatively. Group LD (n=15): Patients will receive same infusion regimen of lidocaine 2%; as in group L plus 0.5 μg/kg dexmedetomidine intravenously as a bolus dose, followed by intravenous infusion of 0.4 μg/kg/h using a 50cc syringe pump intra-operatively. During preoperative visit, evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine, serum electrolytes (sodium, potassium and calcium), fasting blood glucose, liver function tests and any other investigation needed.

* Informed written consent, from all individual participants who will be included in this study will be taken during preoperative visit.
* The patient will be trained during preoperative visit on a visual analogue scale (VAS) for pain, with 0 corresponding to no pain and 10 to the worst pain imaginable.

Pre-anaesthetic preparation and premedication:

* Fasting hours (6 hours to solids and 2 hours for clear fluids).
* Thrombotic prophylaxis (enoxaparin 40 mg) will be started 12 hours before surgery.
* Antiseptic shower will be taken.
* Elastic stockings will be worn.
* Antibiotic prophylaxis: single dose ceftriaxone 2 g intravenously will be given 1 hour before surgical incision according to hospital policy.

On arrival to the operative theater:

* A peripheral cannula (18G) will be inserted in all patients.
* All patients will be premedicated with intravenous (IV) midazolam (0.03 mg.kg-1) shortly before anaesthesia.
* A multichannel monitor (Dräger® Infinity vista XL) will be connected to the patient to display continuous electrocardiography monitoring for heart rate (beat/min) and rhythm, noninvasive arterial blood pressure (NIBP) (mmHg), arterial oxygen saturation (SpO2%) and end-tidal carbon dioxide (ETCO2) (mmHg) and nasopharyngeal core temperature (oC).
* Patients in group L will receive an initial bolus of lidocaine 1.5mg /kg over 10 minutes immediately before the induction of general anaesthesia then 1.5mg/kg/hr lidocaine infusion in a 50cc syringe pump intra- operatively that will be stopped 30 min before end of surgery. The same volume of normal saline 0.9% will be given intravenously over 10 minutes immediately before the induction of anaesthesia then it will be infused using a 50cc syringe pump intra-operatively in the same rate till 30 min before the end of the procedure to assure blinding.
* Patients in group LK will receive same infusion volume of lidocaine as in group L and 0.35 mg/kg bolus over 10 minutes immediately before the induction of general anaesthesia, followed by infusion of 0.2 mg/kg/h of ketamine intraoperatively that will be stopped 30 min before end of surgery.
* Patients in group LD will receive same infusion volume of lidocaine as in group L and bolus infusion of 0.5 μg/kg over 10 min immediately before the induction of general anaesthesia, 0.4 μg/kg/h continuous infusion of dexmedetomidine intraoperatively that will be stopped 30 min before end of surgery.

Anaesthesia:

After giving bolus doeses of the studied drugs, and preoxygenation for 3 minutes, standard anaesthesia will be induced in the three groups with propofol in increments up to 2mg/kg till loss of verbal response, fentanyl 2μg/kg and atracurium 0.5 mg/kg intravenously to facilitate tracheal intubation. Anaesthesia will be maintained with 50% oxygen-air gas mixture and isoflurane 1-1.5 % MAC to maintain adequate depth of anaesthesia. The haemodynamic variables (eg, heart rate or blood pressure) will be maintained within 20% of the preoperative baseline values by adjusting isoflurane concertration and if not patients will be treated with additional boluses of fentanyl 0.5 mcg/kg intraoperatively as needed.. Mechanical ventilation will be performed with a constant tidal volume of 8 ml/ kg and a respiratory rate of 10 to 12 cycles/min to maintain the end-tidal carbon dioxide tension between 35 and 40 mmHg and an oxygen saturation of ≥ 98 per cent with 50 percent oxygen in air. Incremental doses of atracurium 0.1 mg/kg will be given to maintain muscle relaxation according to nerve stimulator. In all groups, If the MAP drop below 60 mmHg, ephedrine 5 mg IV bolus and fluid bolus will be given and repeated if required. Atropine 0.5 mg IV bolus will be given if HR decreases to less than 50 beats/min. All patients will receive a strict fluid replacement according to the standard fluid administration guidelines during anaesthesia.(19)

* Blood transfusion will be considered only when the patient's blood loss reached the transfusion point as illustrated in the following equation,(20) which will be determined preoperatively from the initial hematocrit, by estimating blood volume and the acceptable hematocrit value will be 25%
* Maintain normothermia: (core temperature not less than 36°C) will be done by actively maintained using bair hugger and warm intravenous fluids.
* Urinary catheter will be inserted for monitoring of urine output.
* All the procedures will be performed by expert surgeons with a clinical experience of more than 5 years in pelvi-abdominal cancer surgeries.
* Patient who will require perioperative blood transfusion will be excluded from the study and will be replaced by another patient to keep the number of each group (15).
* At the end of surgery, anaesthesia will be discontinued; residual neuromuscular block will be reversed by atropine 0.02 mg/kg and neostigmine 0.04 mg/kg. Extubation will be performed awake after the return of protective airway reflexes.

Postoperative Management:

* All patients will be transferred to the intermediate care unit and will be closely monitored continuously for the next 24 hours by observers who will be blinded to study groups. In the three groups, intravenous paracetamol 1 g/6 hours (Perfalgan® 100 ml vial UPSA France) will be given for postoperative pain as standard in our institute. Intravenous ketorolac 15 mg/8 hours will be given for postoperative pain relief if VAS is still ≥ 4 as first postoperative rescue analgesic. Fentanyl 0.5 mcg/kg IV will be given as second postoperative rescue analgesic if VAS was ≥ 4 inspite of giving ketolac.
* The incidence of postoperative nausea and vomiting (PONV) will be assessed by a nurse for the first 24 hrs and only 2 possible answers will be accepted (yes or no). Nausea is defined as subjective sensation of discomfort associated with the awareness of the urge to vomit. Vomiting is defined as a forceful expulsion of gastric contents through the mouth. Rescue anti-emetic ondansetron 8 mg intravenously will be given if the patient has persistent nausea or more than a single episode of vomiting or whenever patients request medication.
* Study participants, including patients, attending anesthesiologists, surgeons, and all data collectors, will be all unaware of the drug in each syringe, and the master codes will be held by a person who does not participate in the observation.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years.
* Female patients.
* ASA physical status class I or II.
* Elective resectable pelvi-abdominal cancer.

Exclusion Criteria:

* Patients with history of sensitivity to the studied drugs.
* Patients with cardiac conduction defects.
* Impaired kidney or liver function.
* Psychiatric disease or seizure disorder requiring medication within the previous 2 years.
* Opioid tolerant patient.
* Patient receiving nonsteroidal anti-inflammatory drugs within 1 week of surgery.
* Patient receiving B blockers, α2 ad-renergic agonist, sedatives, and antiarrythemic drugs.
* Cognitive dysfunction.
* Any history of antitumor treatments before surgery.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Serum pro-inflammatory cytokines (IL-1, IL-6, TNFα). | Preoperative, 2 hours after recovery and after 24 hours

SECONDARY OUTCOMES:
• Pulse rate (Beats / min). | Intraoperative
Propofol consumption at induction (mg). | Intraoperative
Post-operative pain score. | Visual analogue scale will be assessed every 2 hours postoperatively for 8 hours then at 12, 18 and 24 hours postoperatively.
  Visual analogue scale
Time to first postoperative analgesic request (min). | First 24 hours
  Time to first postoperative analgesic request (min) which is the time elapsed between end of surgery and first administration of an analgesic.
Perioperative analgesic consumptions. | First 24 hours
  Postoperative Ketolac requirements (mg). Postoperative fentanyl requirements (μg).
Recovery profiles. | Postoperative upto 60 minutes
  Time to spontaneous eye opening defined as time from the end of anaesthesia to eye opening on command (min). Time to extubation defined as time from the end of surgery to tracheal extubation (min). The time at which the patients will attain an Aldrete score >9 in minutes will be recorded.
Length of hospital stay in days. | Upto 14 days after surgery
Adverse effects | First 24 hours
  Example as Incidence of postoperative nausea and vomiting
• Non-invasive measurement of mean arterial blood pressure (in mmHg). | Intraoperative
• Pulse oxygen saturation. (SpO2%) | Intraoperative
Average end tidal concentration of isoflurane (%). | Intraoperative
Intraoperative fentanyl requirements (μg). | Intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Through clinical trials
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months upto 1 year
Access Criteria: Lidocaine, ketamine, dexmedetomidine, pelvi-abdominal cancer, proinflammatory cytokines

REFERENCES:
- [Background] Hassan MM, Saleh RG, Abdalla NO, Radwan NH, Abdelghfar EM. Effect of lidocaine infusion compared to dexmedetomidine infusion on proinflammatory cytokines and stress response in pelvi-abdominal cancer surgeries: a randomized clinical trial. Anaesth. pain intensive care 2021;26 (1):44-52. DOI: 10.35975/apic.v26i1.1765